CLINICAL TRIAL: NCT01409772
Title: Evaluation of the Clinical Practice of Using of a 70 % Ethanol Lock Solution for the Prevention of Catheter Related Blood Stream Infections in Pediatric Patients Undergoing Intestinal Rehabilitation
Brief Title: Evaluation of 70% Ethanol Lock Solution to Prevent Catheter Related Blood Stream Infections in Pediatric Patients
Status: Withdrawn | Type: Observational
Why Stopped: PI decided to withdraw study
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0156-09-FB
Record Dates: First submitted 2009-05-22; First posted 2011-08-04 (Estimated); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Blood Stream Infections; Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome | interventions — Ethanol

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intestinal Rehab: Pediatric Patients Undergoing Intestinal Rehabilitation for short bowel syndrome
  Interventions: Drug: Ethanol Lock

INTERVENTIONS:
Drug: Ethanol Lock — Ethanol Lock
  Other Names: 70% ethanol

SUMMARY:
The purpose of this study is to evaluate the clinical practice of the prophylactic use of ethanol locks for the prevention of catheter related blood stream infections in pediatric intestinal rehabilitation program patients requiring total parenteral nutrition.

DETAILED DESCRIPTION:
Catheter- related blood stream infections are a serious complication for pediatric patients receiving parenteral nutrition. The leading causes of death in infants with short bowel syndrome (SBS) who are being treated with parenteral nutrition are central line sepsis and liver failure associated with the prolonged use of parenteral nutrition. (Cuffari, 2006) Incidence of infection ranges from 3% to 60% over the life span of each catheter. (Fratino, 2002) Interruption of nutritional support, antibiotic resistance and septic complications resulting from frequent infections can be life threatening to this fragile patient population. This patient population is dependent upon maintenance of central venous access for survival. Frequent hospitalizations, loss of work, and financial complications result in decreased quality of life for these patients and their caretakers. The cost of hospital treatment of catheter related bloodstream infections (CRBSI) has been estimated to range from $4000 to $56,000 for each occurrence. (MMWR 2002)

Vascular access sites are also limited in the pediatric population, and removal of central access for infection may diminish future ability to provide vital parenteral nutrition.(MMWR, 2002) Therefore, improvements in the ability to prevent infection are of utmost importance in this patient population.

The concept of antibiotic lock technique was developed in the late 1980s and was derived from various heparin lock protocols. Antibiotic locks have been used for both management and prevention of infection in vascular access devices. Antimicrobial choices for use in the antibiotic lock technique are dependent on the different pathogens suspected to infect the catheter lumen, characteristics of the organisms, and the pharmacodynamic properties of the antimicrobial agent. There is a risk of selection for multi-drug resistant organisms when antibiotic locks are utilized. In addition, heparin must be added to an antibiotic lock solution to maintain catheter patency.

More recently, ethanol locks have been utilized as a treatment option for children with CRBSIs. Ethanol is not only bactericidal and fungicidal in nature but also reveals thrombolytic properties. (Mouw, 2008) The thrombolytic properties eliminate the need for heparin addition to maintain catheter patency. Although utilized as treatment, ethanol is not currently being used for CRBSI prevention at our institution. Along with decreasing the risk of emerging antibiotic resistance, the investigators are attempting to determine if using ethanol as a lock solution will diminish the number of infections in the Intestinal Rehabilitation Program population, leading to decreased patient complications and costs. UNMC has the largest population of Intestinal Rehabilitation Program participants in the country making this a uniquely well-suited clinic in which to gather data surrounding this emerging infection-prevention strategy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent/assent and willingness to adhere to protocol
* Intestinal rehabilitation patients with documented short bowel syndrome
* Age: newborn to 19 years of age
* Indwelling tunneled venous catheter placed for the purpose of total parenteral nutrition/IV fluids, with a 2 hour or longer window out of 24 hours for ethanol lock instillation
* No history of alcohol abuse
* No history of hypersensitivity to ethanol
* No history or documented active seizure disorder

Exclusion Criteria:

* Parent/guardian unwilling to sign consent
* Active bacterial infection
* Non-tunneled, non-permanent catheter (triple lumen or PICC)
* Pre-existing condition that would prevent enrollment as determined by each patients' physician
* Inability to adhere to protocol

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Short Bowel Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-05 (Estimated); Primary Completion 2009-07-09 (Actual); Study Completion 2009-07-09 (Actual)

PRIMARY OUTCOMES:
90 day infection rate prior to enrollment | 90 days
  To determine the 90 day infection rate in eligible subjects for the term immediately prior to enrollment in the study protocol.

SECONDARY OUTCOMES:
90 day CRBSI rate | 90 days
  90 day CRBSI rate in enrolled subjects.
Organism and Treatment in CRBSI | 90 days
  Type of organism involved in CRBSI, and the treatment strategy used for each infection.

CONTACTS AND LOCATIONS:
Overall Officials: Kari A Simonsen, MD, Principal Investigator — UNMC